CLINICAL TRIAL: NCT06901115
Title: Corkscrew Technique: A Novel Modification in Transurethral Resection of Large Prostate (60-100 g) Optimizing Resection Efficacy and Safety: A Double-blind Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ammar Fathi Mohamed AlOrabi, Doctor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Corkscrew technique
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: TURP(Transurethral Resection of Prostate); BPH (Benign Prostatic Hyperplasia); Prostate
Keywords: TURP; BPH; Prostate; Blandy; Nesbit
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nesbit technique group (Sham Comparator): patients of this group undergo the classical Nesbit technique.
  Interventions: Procedure: Nesbit technique
- Corkscrew technique (Active Comparator): patients of this group undergo the novel modified technique.
  Interventions: Procedure: Corkscrew technique

INTERVENTIONS:
Procedure: Nesbit technique — it is composed of development of trough at the right prostatic lobe (at 10 o'clock) from the bladder neck proximally down to a level just above the external urethral sphincter distally, then deepening the trough until the prostatic capsule, performing haemostasias then resection of lateral lobes in halves, upper right, lower right, upper left and at last lower left respectively with haemostasias in-between. Then resection of the median lobe if present. Final haemostasias then ensues before insertion of the triple way catheter with normal saline irrigation.
  Arms: Nesbit technique group
Procedure: Corkscrew technique — the Corkscrew technique was performed by resection starting at 3 o'clock and carried on in a clockwise manner till 3 o'clock again. Prostate was resected from bladder neck downwards to the verumontanum after dividing the gland, imaginary, into 3 zones or thirds, proximal, middle and distal zone. The gland was resected zone by zone in this corkscrew manner. Once the proximal third is resected and hemostasis done, the middle third resection is done in the same manner, The process is repeated for the distal third. Hemostasis was performed instantly.
  Arms: Corkscrew technique

SUMMARY:
Transurethral resection of the prostate (TURP) is still the gold standard for surgical management of enlarged prostate. However, many techniques and minimally invasive procedures are now in the comparative track with Bipolar resection as Laser enucleation.

Multiple drawbacks of Classic TURP problems related to large prostate management as the retreatment after Bipolar resection, another issue that prolonged operative time, Loss of orientation during resection due to rotation of one of the 2 kissing lobe, Bleeding of the 1st lobe resection side make the 2nd lobe resection harder and lengthier, Median lobe resection or bladder neck resection is done at last to avoid sub-trigonal injury. however, due to median lobe obstruction, irrigation is poor during all the resection. length of learning curve, the modification of early median lobe resection carry the risk of sub-trigonal injury.

So, this study is a trial to analyze the effect of new technique in resection of large prostate with good orientation and less time of operation.

ELIGIBILITY:
Inclusion Criteria:

* BPH causing LUTS with prostate volume between 60 and 100 ml (either by TRUS or CT).
* PSA level below 4 ng/ml.
* IPSS score of 10 and above.

Exclusion Criteria:

* previous history of prostatic biopsy.
* previous history of acute urinary retention.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Weight of resected tissue | within one hour postoperatively
  The weight of resected tissue measured in grams using laboratory scale device.
Resection time | the operative time
  Resection time measured in minutes by documenting the time of resection start and time of resection end.
Complication rate | the operative time
  Complication rate is measured by number of complications occurred.

SECONDARY OUTCOMES:
Change in International Prostate symptom score (IPSS) | one month postoperatively
  The change in International Prostate Symptom Score (IPSS) is measured by difference between preoperative and postoperative IPSS. IPSS is measured by IPSS scoring system in form of numbers, where minimum score is 0 representing no symptoms and maximum score is 35 representing the most sever symptoms.
Change in Qmax | One month postoperatively
  The change in IPSS score is measured by difference between preoperative and postoperative Qmax. Qmax (maximum flow rate) is measured using uroflowmetry and measured by ml/sec.
Change in postvoid residual volume | One month postoperatively
  The change in postvoid residual volume is measured by difference between preoperative and postoperative postvoid residual volume. postvoid residual volume is assessed using pelviabdominal ultrasound and measured by centimeter cubic.
Change in hemoglobin level | One day postoperatively
  The change in hemoglobin is measured by difference between preoperative and postoperative hemoglobin level. Hemoglobin level is assessed using Complete Blood Count and measured by g/dl.

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia Faculty of Medicine, Shebin El-Kom, Menoufia, Egypt